CLINICAL TRIAL: NCT05914402
Title: Axillary Surgery De-escalation After Neoadjuvant Therapy (NeoaPET) Using a Dedicated Breast PET-based Pathological Response-adapted Strategy in Patients With Axillary-positive Early Breast Cancer
Brief Title: Axillary Surgery De-escalation After Neoadjuvant Therapy Using Dedicate Breast PET
Acronym: NeoaPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-NeoaPET
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: breast cancer, Neoadjuvant Therapy, Dedicate Breast PET, axillary surgery de-escalation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation group( Axillary surgical evaluation is spared) (Experimental): Breast cancer patients with initial axillary metastasis（T1-3N1-3M0） who are preparing for neoadjuvant therapy(NAT)，including neoadjuvant chemotherapy, targeted therapy, immunotherapy, etc. will received imaging examination（MRI、mammography、ultrasonography）at baseline and after every two cycles of NAT before surgery, dedicated breast/lymph positron emission tomography(DB/L-PET) at baseline and after first 1-2 cycle of NAT. We have developed a prediction model, which includes clinical parameters, pathological parameters, imaging examination parameters and DB/L-PET to predict the probability of complete pathological remission of axillary lymph nodes after receiving NAT. If the probability is more than 90%, the process of axillary surgical evaluation will be spared. If the probability is 50% -90%, Sentinel lymph node biopsy will be performed. If the probability is less than 50%, standard axillary lymph node dissection will be performed.
  Interventions: Procedure: axillary surgery de-escalation after NAT

INTERVENTIONS:
Procedure: axillary surgery de-escalation after NAT — the process of axillary surgical evaluation will be spared after NAT using the prediction model if the probability is more than 90%.

SUMMARY:
Some breast cancer patients with initial axillary metastasis can achieve axillary complete pathological remission(A-pCR) after neoadjuvant therapy(NAT)，These patients are candidates for axillary Surgery de-escalation. This prospective study is designed to evaluate the feasibility and safety of axillary surgery de-escalation for the initial axillary metastasis breast cancer patients who are predicted to achieve A-pCR using multiple pathological indicators and imaging examinations (molecular typing, ultrasound and dedicated breast positron emission tomography, etc.) before and after 1-2 cycles NAT

ELIGIBILITY:
1. Clinical stage T1-3 N1-3M0 breast cancer at diagnosis (prior to neoadjuvant chemotherapy) by American Joint Committee on Cancer (AJCC) staging 8th edition 2. No inflammatory breast cancer 3. No other malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix 4. All patients must have had an axillary ultrasound with fine needle aspiration (FNA) or core needle biopsy (CNB) of axillary lymph nodes documenting axillary metastasis at the time of diagnosis, prior to or at most 14 days after starting neoadjuvant chemotherapy (NAC)

* Note: Biopsy of intramammary nodes does not fulfill eligibility criteria; In some patients, a clip is implanted into positive lymph nodes verified by FNA or CNB under the guidance of ultrasound 5. Patients must have had estrogen receptor, progesterone receptor and HER2 status (by immunohistochemistry [IHC] and/or in situ hybridization [ISH]) evaluated on CNB prior to start of NAC 6. Patients must have completed all planned cycles and regimens of NAC prior to surgery; patients must have completed at least 4 cycles of NAC consisting of an anthracycline and/or taxane-based regimen without evidence of disease progression in the breast or the lymph nodes
* Note: Delays/dose modifications due to toxicities/adverse events are allowed as long as a minimum of 4 cycles of NAC is administered; more than 4 cycles of NAC may be administered at the discretion of the treating medical oncologist 7. Patients with HER-2 positive tumors must have received neoadjuvant trastuzumab, or trastuzumab + pertuzumab, or other approved anti-HER-2 therapy (either with all or with a portion of the NAC regimen); therapy must be Food and Drug Administration (FDA)-approved targeted anti-HER2 therapy, but additional therapies are allowed as are non-trastuzumab regimens if administered in the context of an Institutional Review Board (IRB)-approved clinical trial 8. All patients must have a clinically negative axilla (no bulky adenopathy) on physical examination documented at the completion of NAC
* Note: an ultrasound of the axilla is not required at completion of NAC; if performed, its findings do NOT impact eligibility 9. No more than 8 weeks of neoadjuvant endocrine therapy prior to the start of NAC 10. No neoadjuvant radiation therapy 11. No SLN surgery/excisional biopsy for pathological confirmation of axillary status prior to or during NAC 12. No prior history of ipsilateral breast cancer (invasive disease or ductal carcinoma in situ [DCIS]); lobular carcinoma in situ (LCIS) and benign breast disease is allowed 13. No prior ipsilateral axillary surgery, such as excisional biopsy of lymph node(s) or treatment of hidradenitis 14. No history of prior or concurrent contralateral invasive breast cancer; benign breast disease; LCIS or DCIS of contralateral breast is allowed 15. Patients must not be pregnant or nursing
* Note: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential 16. Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1 16. Patients must have completed first dedicated breast PET (dbPET) at baseline before starting NAC, and can be expected to undergo second dedicated breast PET before second or third cycle NAC.

  17. We have designed a calculation model (including various clinical, pathological, imaging, and imaging omics indicators, especially dbPET) where patients who meet the model's calculation results are exempt from axillary surgical evaluation, while those who do not meet the model's calculation results are treated with standard axillary surgical treatment based on the patient's axillary condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-18 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Node Recurrence Rate | 2 years
  a recurrence in the ipsilateral axillary, supraclavicular, or internalmammary nodal basins.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No